CLINICAL TRIAL: NCT02247362
Title: Phase 1b/2 Double Blind, Randomized, Placebo Controlled Study of Safety and Immunogenicity of VAX2012Q: A Quadrivalent Influenza Vaccine in Healthy Adults Age 65-75 Years
Brief Title: Study of Safety and Immunogenicity of a Quadrivalent Influenza Vaccine in Healthy Adults Age 65-75 Years
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAX2012Q-02
Record Dates: First submitted 2014-09-18; First posted 2014-09-25 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: Safety; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vaccine Dose Group 12 mcg (Experimental): VAX2012Q, 12 mcg dose
  Interventions: Biological: VAX2012Q
- Vaccine Dose Group 20 mcg (Experimental): VAX2012Q, 20 mcg dose
  Interventions: Biological: VAX2012Q
- Vaccine Dose Group 16 mcg (Experimental): VAX2012Q; 16 mcg dose
  Interventions: Biological: VAX2012Q
- Vaccine Diluent (Placebo Comparator): Vaccine Diluent, F147, as placebo control
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: VAX2012Q — Recombinant influenza HA vaccine consisting of two Influenza A subtypes and two Influenza B lineages and delivered IM
  Other Names: Quadrivalent Recombinant Hemagglutinin Influenza Vaccine
  Arms: Vaccine Dose Group 12 mcg; Vaccine Dose Group 16 mcg; Vaccine Dose Group 20 mcg
Other: Placebo — Vaccine Diluent
  Other Names: Vaccine Diluent
  Arms: Vaccine Diluent

SUMMARY:
One dose of escalating strengths of an investigational influenza vaccine, VAX2012Q (Quadrivalent Recombinant Hemagglutinin Seasonal Influenza Vaccine), will be evaluated for safety and immunogenicity in healthy adults 65 to 75 years of age in this placebo-controlled study.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate, in a stepwise fashion, dose levels for an investigational quadrivalent influenza vaccine containing 2 influenza A strains and 2 influenza B strains. This is a multi-center, randomized, double-blind, placebo-controlled, dose escalating study in which up to 200 healthy adults age 65-75 years will be administered a single dose of either placebo or an investigational influenza vaccine (VAX2012Q, Quadrivalent Recombinant Hemagglutinin Seasonal Influenza Vaccine) at one of up to 3 dose levels. Fifty or up to 75 subjects will be enrolled in each dose level. Data for safety and immunogenicity will be collected for all dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 65-75 years of age at the time of vaccination in good health. Individuals that are stably treated for hypertension may be eligible.
* Able to provide informed consent
* Willing to receive the unlicensed vaccine
* Willing to provide multiple blood specimens
* Live in the community, independently or in an assisted living environment
* Based on the results of the Short Portable Mental Status Questionnaire be rated as normal or have no greater than mild severity dementia
* As defined by the Canadian Study of Health and Aging Clinical Frailty Scale be a Class 1 to 5

Exclusion Criteria:

* Preceding the administration of study vaccine, has received or will receive 1) any licensed or investigational influenza vaccine product within 6 months, 2) any investigational drug or any investigational vaccine product other than influenza vaccine within the 30 days, 3) any licensed live vaccine other than influenza vaccine within 4 weeks, 4) any licensed inactivated vaccine other than influenza vaccine within 2 weeks
* Planned receipt before the Day 21 blood draw of 1) any licensed or investigational influenza vaccine product, 2) any investigational drug or any investigational vaccine product other than influenza vaccine, 3) any licensed live vaccine other than influenza vaccine, 4) any licensed inactivated vaccine other than influenza vaccine
* History of excessive alcohol use, drug abuse or significant psychiatric illness
* Has a chronic illness that is not medically stable, is receiving a concomitant therapy in which the medication dose has not been stable for at least 3 weeks prior to immunization or has any other condition that could interfere with the subject's participation in the study or interpretation of the study results
* Clinically significant abnormal liver function tests at screening
* Subjects with Grade 2 or higher abnormalities in total bilirubin at screening
* Subjects with any of the following laboratory abnormalities at screening: Creatinine >1.7mg/dL, Hemoglobin < 11g/dL for females; <12.5 g/dL for males, WBC <2500cell/mm3 or > 15,000cell/mm3 and Platelet Count <125,000cell/mm3
* Positive serology of HBSAg, HCV or HIV antibodies
* Having cancer or have received treatment for cancer within three years, excluding minor skin cancers, which are allowed unless located at the vaccination site. Persons with a history of cancer who are disease-free without treatment for three years or more are eligible.
* Persons with impaired immune responsiveness (of any cause), including Type 1 diabetes mellitus and auto immune disorders or any known or suspected autoimmune disease
* Persons with congenital immunodeficiency or history of acquired immunodeficiency, or immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding six months.
* Persons with a history of severe allergic reaction after previous vaccinations or hypersensitivity to any seasonal influenza vaccine component
* Persons with a history of Guillain-Barré Syndrome
* Receipt or donation of blood or blood products 8 weeks prior to vaccination or during the three week study period following vaccination
* Acute disease within 72 hours prior to vaccination.
* An oral temperature >100.4°F (38°C)
* Systolic blood pressure < 85 mm Hg and subjects whose hypertension is untreated or unstable with antihypertensive therapy or that have systolic BP ≥ 160 mm Hg or diastolic BP ≥ 100 mm Hg requiring medical intervention with more than one drug or more intensive therapy than previously used or indicated.
* Body Mass Index >40
* Disorders of coagulation
* Women less than 1 year post menopausal
* A clinical diagnosis of influenza within the previous 6 months
* Any other condition or circumstance which, in the opinion of the Principal Investigator, poses an unacceptable risk for participation in the study

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Injection site and systemic symptoms will be collected for 21 days after vaccination. Other AEs assessed as related to vaccination will be collected at a 6 month and 1 year phone call. | 21 days post-immunization; follow up at 6 months and one year

SECONDARY OUTCOMES:
Immune response to vaccine will be measured by serum HAI levels | 21 days post-immunization

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Tussey, PHD, Study Director — VaxInnate Corporation
Locations (3):
- Australia (3):
  - Q-Pharm Pty Limited, Herston, Queensland
  - CMAX, a division of IDT Australia Limited, Adelaide, South Australia
  - Linear Clinical Research Limited, Nedlands, Western Australia